CLINICAL TRIAL: NCT04601168
Title: Assessment of the Safety and Performance of a Compression Knee Support in the Prevention of Injuries During Sports Practice
Status: Terminated | Type: Observational
Why Stopped: Difficulties of inclusion, financial considerations, review of CER (no additional clinical data needed to demonstrate safety and performance of the medical device under evaluation)
Sponsor: Decathlon SE (Industry)
Collaborators: EFOR, France (Industry)
Responsible Party: Sponsor
Other Study IDs: kneeSOFT100
Record Dates: First submitted 2020-09-04; First posted 2020-10-23 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Chronic Knee Pain; Chronic Instability of Knee Joint

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: kneeSOFT100 — During the first two weeks of follow-up, the subject shall not use the device during the sports sessions. The subject shall use the device during the sports sessions for the next 4 weeks (6 weeks of follow-up)

SUMMARY:
Decathlon has developed kneeSOFT100 product which is medical device designed to reduce pain and joint instability during sport practice. The objective of this multicentre study is to collect data on the related clinical complications and clinical outcomes of market-approved Decathlon kneeSOFT100 product to demonstrate safety and performance of this device in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Subject is aged ≥18 years old
* Subject has chronic pain AND / OR chronic knee instability
* The current condition of his/her knee allows the subject to resume usual physical activity
* Subject has been informed and is willing to sign an informed consent form
* Subject is willing to comply with protocol requirements and return to the study center for all clinical evaluations and required follow-up (6 weeks)
* Subject is affiliated to the French social security regime

Exclusion Criteria:

* Subject has conditions that may interfere with his/her ability to understand protocol requirements, participate in scheduled visits, or provide his/her informed consent
* Subject has worn a support (knee brace or articulated orthosis) during sports sessions during the last month
* Subject has any medical condition that could impact the study at investigator's discretion
* Subject has a known hypersensitivity or allergy to the components of the device (elastodiene, polyester)
* Adult subject to a legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject with chronic pain AND / OR chronic knee instability whose current condition of his/her knee allows him/her to pursue a usual physical activity.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Functional score | 6 weeks of follow-up
  Comparison of the functional result (Lysholm Score: 0-100 points) between the baseline and last follow-up visit

SECONDARY OUTCOMES:
Confidence level | At baseline and 6 weeks of follow-up
  Gap in the confidence level (patient rated outcome with 6 questions, ranging from 0 to 100) related to physical activity, between the baseline and last follow-up visit
Knee instability | At 2 weeks and 6 weeks of follow-up
  Comparison of knee instability between the first two weeks of follow-up (without use of the device during sports sessions) and the following four weeks (with use of the device during sports sessions), measured through a numerical rating scale (NRS, ranging from 0 to 10)
Knee pain | At 2 weeks and 6 weeks of follow-up
  Comparison of knee pain between the first two weeks of follow-up (without use of the device during sports sessions) and the following four weeks (with use of the device during sports sessions), measured through a NRS (ranging from 0 to 10)
Safety (adverse events) | 6 weeks of follow-up
  Rate of adverse events occurred during the study

CONTACTS AND LOCATIONS:
Overall Officials: Valérie WIECZOREK, Principal Investigator — Centre Hospitalier Universitaire de Lille
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire de Lille, Lille
  - KOSS Paris 8, Paris